CLINICAL TRIAL: NCT05787106
Title: Role of Adverse Childhood Events and Rejection Sensitivity on Alcohol Use in Recently Withdrawn Individuals With Alcohol Use Disorder
Acronym: TRAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2022-2/AL-01
Record Dates: First submitted 2023-03-13; First posted 2023-03-28 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Alcohol-Induced Disorders; Ostracism
Keywords: Adverse childhood experiences; Rejection
MeSH Terms: conditions — Alcohol-Induced Disorders; Ostracism; Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PAtients withdrawn from alcohol (Experimental)
  Interventions: Other: Cyberball task

INTERVENTIONS:
Other: Cyberball task — The game consists of ball throws between animated characters lasting about 50 throws. In the rejection condition, after 2 or 3 throws, the participant no longer receives the ball (no more passes). In the control conditions ("all included"), the participant receives the ball as often as the others.

SUMMARY:
Low utilization of addiction treatment is a public health problem. A number of factors are associated with lack of treatment, including public stigma, self-stigma, and beliefs that people with addiction should solve their problem on their own. Stigma exposes individuals to social rejection, which may sustain the anxiety of rejection, and exacerbate certain mental disorders such as addictions. Social cognition disorders have been shown to be present in addictions, but one dimension of social cognition, emotional sensitivity to rejection (ESR), has been less studied. Rejection sensitivity could be considered a critical element in access to care and the relapse process.

The study authors hypothesize a role for emotional dysregulation in rejection situations in the relapse of alcohol use disorder in recently withdrawn patients. Specifically, they hypothesize that participants with a greater change in negative experience after a rejection situation on a Cyberball task, as measured by the negative subscale of the Positive and Negative Affect Schedule (PANAS), will have a higher percentage of days with heavy drinking during the last four weeks to three months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the Grau-du-Roi Follow-up and Rehabilitation Care Service.
* Patient abstinent from alcohol for at least 10 days.
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* Other mental health disorder: bipolar disorder, schizophrenia, severe acute depression, borderline personality.
* Severe substance use disorder (SUD).
* Current suicidal ideation as judged by clinician.
* Patient unable to give consent.
* Pregnant or breastfeeding patient.
* The subject is participating in a Category 1 interventional study, or is in a period of exclusion determined by a previous study
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Role of emotional reaction to social rejection (Cyberball game) | Day 0; before Cyberball task
  Positive And Negative Affect Schedule (PANAS) (negative affect score). Scores can range from 10 to 50 for positive and negative emotions, with lower scores representing lower levels of positive/negative emotional engagement and higher scores representing higher levels of positive/negative emotional engagement.
Role of emotional reaction to social rejection (Cyberball game) | Day 0; after Cyberball task
  Positive And Negative Affect Schedule (PANAS) (negative affect score). Scores can range from 10 to 50 for positive and negative emotions, with lower scores representing lower levels of positive/negative emotional engagement and higher scores representing higher levels of positive/negative emotional engagement.
Percentage of heavy drinking days in the past 4 weeks | Month 3
  Timeline Follow Back (TLFB) interview
Correlation between percentage of heavy drinking days and the difference between the PANAS negative subscale scores at baseline and after the Cyberball task in the exclusion phase (=rejection situation). | Day 0; before Cyberball task
  Multiple linear regression
Correlation between percentage of heavy drinking days and the difference between the PANAS negative subscale scores at baseline and after the Cyberball task in the exclusion phase (=rejection situation). | Day 0; after Cyberball task
  Multiple linear regression
Correlation between percentage of heavy drinking days and the difference between the PANAS negative subscale scores at baseline and after the Cyberball task in the exclusion phase (=rejection situation). | Month 3
  Multiple linear regression

SECONDARY OUTCOMES:
Adverse childhood events | Day 0
  Adverse childhood events (ACE) score
Patient level of distress due to rejection | Day 0; after Cyberball task
  Need Threat Scale (NTS) score
Patient self-stigma due to alcohol dependence | Day 0
  Self-stigma in Alcohol Dependence (SSAD) scale score
Patient depression | Day 0
  Patient Health Questionnaire (PHQ-9) score
Patient depression | Month 3
  Patient Health Questionnaire (PHQ-9) score
Patient depression | Month 6
  Patient Health Questionnaire (PHQ-9) score
Patient depression | Month 12
  Patient Health Questionnaire (PHQ-9) score
Patient anxiety | Day 0
  Generalized Anxiety Disorder-7 (GAD-7) score
Patient anxiety | Month 3
  Generalized Anxiety Disorder-7 (GAD-7) score
Patient anxiety | Month 6
  Generalized Anxiety Disorder-7 (GAD-7) score
Patient anxiety | Month 12
  Generalized Anxiety Disorder-7 (GAD-7) score
Number of days of alcohol consumption in the past 4 weeks | Month 3
  Timeline Follow Back (TLFB) interview
Number of days of alcohol consumption in the past 4 weeks | Month 6
  Timeline Follow Back (TLFB) interview
Number of days of alcohol consumption in the past 4 weeks | Month 12
  Timeline Follow Back (TLFB) interview
Number of days of heavy alcohol consumption in the past 4 weeks | Month 3
  Timeline Follow Back (TLFB) interview
Number of days of heavy alcohol consumption in the past 4 weeks | Month 6
  Timeline Follow Back (TLFB) interview
Number of days of heavy alcohol consumption in the past 4 weeks | Month 12
  Timeline Follow Back (TLFB) interview
Percentage of heavy drinking days in the past 4 weeks | Month 3
  Timeline Follow Back (TLFB) interview
Percentage of heavy drinking days in the past 4 weeks | Month 6
  Timeline Follow Back (TLFB) interview
Percentage of heavy drinking days in the past 4 weeks | Month 12
  Timeline Follow Back (TLFB) interview
Lifetime history of suicide attempts | Day 0
  Number
Current treatments | Day 0
  List of current treatments taken from patient medical file
Patient dispositional (i.e. trait) empathy | Day 0
  Interpersonal reactivity index (IRI) score
Concurrent validity of the Adult rejection Sensitivity Questionnaire (A-RSQ) with the Positive And Negative Affect Schedule (PANAS) after the rejection situation. | Day 0; before Cyberball task
Concurrent validity of the Adult rejection Sensitivity Questionnaire (A-RSQ) with the Positive And Negative Affect Schedule (PANAS) after the rejection situation. | Day 0; after Cyberball task
Concurrent validity of the Adult rejection Sensitivity Questionnaire (A-RSQ) with the Need Threat Scale (NTS) after the rejection situation. | Day 0; before Cyberball task
Concurrent validity of the Adult rejection Sensitivity Questionnaire (A-RSQ) with the Need Threat Scale (NTS) after the rejection situation. | Day 0; after Cyberball task

CONTACTS AND LOCATIONS:
Overall Officials: Amandine Luquiens, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No